CLINICAL TRIAL: NCT05076968
Title: Association Between Patient Satisfaction With Complete Dentures and the Clinical Experience of the Treating Dentist
Brief Title: Patient Satisfaction and Clinical Experience of Dentists
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Dr. Nadia Ereifej, AssociateProfessor, University of Jordan
Other Study IDs: YOweis
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Patient Satisfaction
Keywords: Complete denture; Patient satisfaction; survey; edentulous patients; treatment outcomes
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Complete dentures fabricated by undergraduate students
  Interventions: Procedure: Complete denture fabrication
- Complete dentures fabricated by prosthodontists
  Interventions: Procedure: Complete denture fabrication

INTERVENTIONS:
Procedure: Complete denture fabrication — Patient satisfaction was assessed regarding dentures fabricated by students and specialists after 8 weeks of delivery

SUMMARY:
Rehabilitation of the edentulous patients has always been a challenge. The success of this treatment modality is not only affected by the patients' acceptance of his new dentures, but on his ability to use them which depends to a great extent on the quality of those dentures. It is strongly believed that the success of dental treatments is affected by the experience of a dentist. The aim of this study was to compare patient satisfaction with complete dentures provided by forth and fifth year dental students and prosthodontists at the University of Jordan Hospital one week and 8 weeks post insertion

DETAILED DESCRIPTION:
After obtaining the ethical approval, questionnaires were distributed to a total of 60 patients who accepted to participate in this study. The 60 patients consisted of 2 groups. The first group included patients treated by fourth and fifth year students, the second group consisted of patients treated by prosthodontists with a minimum of 5 years of experience. The questionnaire was distributed to those patients 8 weeks post insertion of complete upper and lower dentures. The questionnaire was divided into 3 parts. the first part included demographic and contact information questions for the patient. The second part included examination to the upper and lower dental arches and a third part included questions that probed the patient's satisfaction with his upper and lower dentures in general. Furthermore, the questionnaire included questions about the patient's comfort with his dentures, whether he is satisfied with the esthetics, phonetics, retention, efficiency in mastication, and ease of cleaning. This part of the survey was adapted from the Oral Health Impact Profile (OHIP-EDENT) questionnaire.

ELIGIBILITY:
Inclusion Criteria:The study population was completely edentulous patients attending the undergraduate students' clinic and specialty Prosthodontic clinics at the Jordan University Hospital in need of conventional complete dentures.

-

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population was completely edentulous patients attending the undergraduate students' clinic and specialty Prosthodontic clinics at the Jordan University Hospital in need of conventional complete dentures.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 8 weeks after delivery
  Visual Analogue Scale based questionnaire with 10 items regarding patient satisfaction
OHIP-EDENT | 8 weeks after delivery
  20 item questionnaire regarding the oral health impact profile

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No